CLINICAL TRIAL: NCT04216576
Title: Oral Self-Management of Palbociclib (Ibrance®) Using Mobile Technology
Brief Title: A Study of the Use of Text Message Reminders to Take Palbociclib
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-458
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Palbociclib; Memorial Sloan Kettering Cancer Center; 19-458
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Participants will have a diagnosis of breast cancer and will be taking Palbociclib. Participants will receive standard of care
  Interventions: Other: Paper Drug Diary
- Standard of Care + Intervention (Experimental): Participants will have a diagnosis of breast cancer and will be taking Palbociclib. Participants will receive standard of care + unidirectional text messaging intervention
  Interventions: Other: OhMD APP

INTERVENTIONS:
Other: Paper Drug Diary — Participants will receive and use a paper Drug Diary and a paper medication calendar.
  Arms: Standard of Care
Other: OhMD APP — Participants will receive multiple text messages regarding administration over time on medication self-management over the course of 3 cycles of medication
  Other Names: Unidirectional text messaging
  Arms: Standard of Care + Intervention

SUMMARY:
The purpose of this study is to find out whether it is feasible (acceptable to participants) to use a smartphone app to send text message reminders to take palbociclib, and whether these reminders are effective at helping people remember to take palbociclib according to the treatment schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a breast cancer diagnosis who are initiating therapy on palbociclib (Ibrance)
* >/= 18 years of age
* Able to speak, read and write English
* Willingness and ability to send and receive text messages with intervention app
* Own a mobile telephone "smartphone" with text messaging capabilities. Only iPhone or Android operating systems support OhMD Application
* Criteria applicable for both Control and Intervention groups
* Flip-phones do not support OhMD Application and thus ineligible to participate
* Initiation palbociclib (Ibrance) for the first time, either as monotherapy or in conjunction with other medication such as Lstrozole (Femara) or Fulvestrant (Faslodex)

Exclusion Criteria:

* History of taking palbociclib (Ibrance)
* Patients whose caregivers coordinate their health care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate of medication self-administration | Up to 1 year
  The effectiveness of a mobile technology intervention by calculating the proportion of the number of days that the participant accurately self-administers the medication divided by the number of days the medication should have been taken

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Barton-Burke, PhD, RN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Mazzella-Ebstein A, Barton-Burke M, Anthony V, White C, Zhang Z, Smith A, Robson M. Oral self-management of palbociclib using mobile technology: Findings from a nurse-led randomized controlled trial. Asia Pac J Oncol Nurs. 2024 Oct 15;11(12):100604. doi: 10.1016/j.apjon.2024.100604. eCollection 2024 Dec. PMID 39697813
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org